CLINICAL TRIAL: NCT05673928
Title: A Phase II Study of Tucatinib and Ado-trastuzumab Emtansine (T-DM1) in Patients With HER2-positive Metastatic Solid Tumors and Metastases to Brain (TUCATEMEB)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0899; NCI-2022-11157 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Solid Tumor; Brain Metastases
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Ado-Trastuzumab Emtansine; tucatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tucatinib and Adotrastuzumab Emtansine (T-DM1) (Experimental): Each study cycle is 21 days (3 weeks)
  Participants will take tablets of tucatinib two (2) times a day, about 8-12 hours apart. Participants will receive T-DM1 by vein over about 30 minutes on Day 1 of each cycle
  Interventions: Drug: Trastuzumab emtansine; Drug: Tucatinib

INTERVENTIONS:
Drug: Trastuzumab emtansine — Given by IV (vein)
  Other Names: T-DM1; Trastuzumab-MCC-DM1; Kadcyla; ado-trastuzumab emtansine
Drug: Tucatinib — Given by PO
  Other Names: ARRY-380; ONT-380

SUMMARY:
To learn if the study drugs, tucatinib and adotrastuzumab emtansine (T-DM1), can help to control solid tumors that have spread to the brain.

DETAILED DESCRIPTION:
Primary Objectives:

● To determine the intracranial antitumor activity of the tucatinib and ado-trastuzumab emtansine (T- bination per the modified Response Evaluation Criteria in Solid Tumors (mRECIST) in patients with huma

Key Secondary Objectives:

* To determine the intracranial antitumor activity of the tucatinib and T-DM1 combination per the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria in patients with HER2-positive metastatic solid tumors and brain metastases.
* To evaluate the duration of intracranial response of the tucatinib and T-DM1 combination in patients with HER2-positive metastatic solid tumors and brain metastases.

Other Secondary Objectives:

* To evaluate the safety and tolerability of the tucatinib and T-DM1 combination in patients with HER2-positive metastatic solid tumors and brain metastases.
* To evaluate the systemic antitumor activity of the tucatinib and T-DM1 combination per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 in patients with HER2-positive metastatic solid tumors and brain metastases.
* To evaluate progression-free survival (PFS) in patients with HER2-positive metastatic solid tumors and brain metastases receiving the tucatinib and T-DM1 combination.
* To evaluate overall survival (OS) in patients with HER2-positive metastatic solid tumors and brain metastases receiving the tucatinib and T-DM1 combination.
* To evaluate the duration of response to the tucatinib and T-DM1 combination per the RECIST v1.1 in patients with HER2-positive metastatic solid tumors and brain metastases.
* To evaluate the clinical benefit rate of the tucatinib and T-DM1 combination per the RECIST v1.1 in patients with HER2-positive metastatic solid tumors and brain metastases.

Exploratory Objectives:

* To assess the effects of the tucatinib and T-DM1 combination on cell proliferation and apoptosis.
* To evaluate predictive and pharmacodynamic (PD) biomarkers of response and resistance to the tucatinib and T-DM1 combination.
* To assess the effects of the tucatinib and T-DM1 combination on circulating-free DNA (cfDNA) dynamics.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed HER2-positive metastatic solid tumor. HER2 positivity defined as HER2 overexpression by immunohistochemistry (IHC) 3+ or 2+ and fluorescence in situ hybridization (FISH) positive and/or HER2 amplification by in situ hybridization (ISH) or next generation sequencing (NGS) and/or activating ERBB2 mutation(s) (verified by MDACC Precision Oncology Decision Support).
2. Patients must have one of the following on the screening brain MRI:

   * Untreated brain metastases not requiring immediate local CNS therapy
   * Previously treated brain metastases with progression of previous lesions or new lesions, but not requiring immediate local CNS therapy
   * At least one measurable untreated brain lesion ≥0.5 cm and <3.0 cm in the longest axis
   * Prior SRS radiosurgery (must be completed within 7 days of study treatment initiation) is allowed as long as the previous treatment volume does not overlap with the current targets.
3. Measurable (per the RECIST v1.1) or evaluable extracranial disease.
4. Prior treatment with HER2-targeted treatments such as trastuzumab, pertuzumab, T-DM1, neratinib, lapatinib, or tucatinib is allowed, but not required. Patients with breast and gastric cancer must have received at least 1 line of HER2 targeted treatment.
5. Age ≥18 years at the time of consent.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (Appendix B).
7. Life expectancy ≥3 months, in the opinion of the investigator.
8. Adequate hematological and end-organ function, defined by the following laboratory test results, obtained within 28 days prior to study treatment initiation:

   * Absolute neutrophil count ≥1,200/μL
   * Platelet count ≥100,000/μL
   * Hemoglobin ≥9g/dL
   * Total bilirubin ≤1.5 × upper limit of normal (ULN), except for patients with known Gilbert's disease, who may enroll if conjugated bilirubin is ≤1.5 × ULN
   * Transaminases (AST/ALT) ≤1.5 × ULN (≤5 × ULN if liver metastases are present)
   * Creatinine level <1.5 x ULN or estimated glomerular filtration rate (GFR) ≥50 mL/min/1.73 m2 using the Modification of Diet in Renal Disease (MDRD) study equation as applicable.
9. International normalized ratio (INR) and partial thromboplastin time (PTT)/activated partial thromboplastin time (aPTT) ≤1.5 × ULN, unless on medication known to alter INR and PTT/aPTT. Proprietary Information of MD Anderson Protocol 2021-0899 v.5.0,04/24/2023 28
10. LVEF ≥50% as assessed by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan documented within 3weeks prior to study treatment initiation.
11. For patients of childbearing potential, as defined in Section 4.3, the following stipulations apply:

    * Must have a negative serum or urine pregnancy test (minimum sensitivity of 25 mIU/mL or equivalent units of beta-human chorionic gonadotropin [β-hCG]) result within 3 days prior to study treatment initiation. A patient with a false positive result and documented verification that the patient is not pregnant will be eligible.
    * Must agree not to try to become pregnant during the study and for at least 7 months after the final dose of study treatment
    * Must agree not to breastfeed or donate ova starting at the time of informed consent and continuing through the study and for 7 months after the final dose of study treatment
    * If sexually active in a way that could lead to pregnancy, must consistently use highly effective methods of birth control (i.e., methods that achieve a failure rate of <1% per year when used consistently and correctly) starting at the time of informed consent and continuing throughout the study and for at least 7 months after the final dose of study treatment.

    Highly effective methods of birth control include:

    i. Intrauterine device ii. Bilateral tubal occlusion/ligation iii. Vasectomized partner iv. Sexual abstinence when it is the preferred and usual lifestyle choice of the patient.
12. For patients who can father children, the following stipulations apply:

    * Must agree not to donate sperm starting at the time of informed consent and continuing throughout the study and for at least 7 months after the final dose of study treatment
    * If sexually active with a person of childbearing potential in a way that could lead to pregnancy, must consistently use a barrier method of birth control starting at the time of informed consent and continuing throughout the study and for at least 7 months after the final dose of study treatment
    * If sexually active with a person who is pregnant or breastfeeding, must consistently use a barrier method of birth control starting at the time of informed consent and continuing throughout the study and for at least 7 months after the final dose of study treatment.
13. The patient must provide written informed consent.
14. Must be willing to undergo biopsy as required by the study, if clinically considered safe and feasible by the investigator.

Exclusion Criteria:

1. Patients must not have any of the following on the screening brain MRI:

   * Any untreated brain lesions >3.0 cm in size
   * Any brain lesion thought to require immediate local therapy, including (but not limited to) a lesion in an anatomic site where increase in size or possible treatment-related edema may pose risk to the patient (e.g., brainstem lesions). Patients who undergo local treatment for such lesions may still be eligible for the study based on inclusion criteria #2.
2. Ongoing use of systemic corticosteroids for control of symptoms of brain metastases at a total daily dose of >4 mg of dexamethasone (or equivalent).
3. Poorly controlled (>1/week) generalized or complex partial seizures, or manifestation of neurologic progression due to brain metastases notwithstanding CNS-directed therapy.
4. History of allergic reactions to trastuzumab or compounds chemically or biologically similar to tucatinib, except for Grade 1 or 2 IRRs to trastuzumab that were successfully managed, or known allergy to any of the excipients in the study drugs.
5. Treatment with any systemic anticancer therapy or investigational agent within 5 half-lives (of the drug) or within 21 days (whichever is shorter ) prior to study treatment initiation.
6. Any toxicity related to prior cancer therapies that has not resolved to ≤ Grade 1, with the following exceptions:

   * Alopecia;
   * Neuropathy, which must have resolved to ≤ Grade 2;
   * Congestive heart failure (CHF), which must have been ≤ Grade 1 in severity at the time of occurrence and must have resolved completely.
7. Clinically significant cardiopulmonary disease such as:

   * Ventricular arrhythmia requiring therapy
   * Symptomatic hypertension or uncontrolled asymptomatic hypertension as determined by the investigator
   * Any history of symptomatic CHF, left ventricular systolic dysfunction, or decrease in LVEF
   * Severe dyspnea at rest (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] ≥ Grade 3) due to complications of advanced malignancy or hypoxia requiring supplementary oxygen therapy
   * Grade 2 or greater corrected QT interval (QTc) prolongation on screening electrocardiogram (ECG).
8. Known myocardial infarction or unstable angina within 6 months prior to study treatment initiation.
9. Unable for any reason to undergo contrast MRI of the brain.
10. Have used a strong cytochrome P450 (CYP)2C8 inhibitor within 5 half-lives of the inhibitor, or a strong CYP3A4 or CYP2C8 inducer within 5 days prior to study treatment initiation. Concomitant use of strong CYP3A4 inducers or CYP2C8 inducers or inhibitors is also prohibited during study treatment and for 2 weeks after discontinuation of study treatment. Use Proprietary Information of MD Anderson of sensitive CYP3A substrates should be avoided 2 weeks prior to study treatment initiation and during study treatment.
11. Known carrier of hepatitis B or hepatitis C virus or has other known chronic liver disease.
12. Known positive human immunodeficiency virus status.
13. Patients who are pregnant, breastfeeding, or planning to become pregnant from the time of informed consent until 7 months after the last dose of study treatment.
14. Unable to swallow pills or has significant GI disease that would preclude adequate oral absorption of medication.
15. Other medical, social, or psychosocial factors that, in the opinion of the investigator, could impact patient safety or compliance with study procedures.
16. Evidence within 1 year of the start of study treatment of another malignancy that required systemic treatment.
17. Patients who are eligible for the HER2CLIMB-02 study (NCT03975647) and they can be enrolled in that study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Ecaterina Dumbrava, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org